CLINICAL TRIAL: NCT01413594
Title: Randomized Clinical Trial of Hand Arm Bimanual Intensive Therapy (HABIT)
Brief Title: Bimanual Training in Children With Hemiplegia
Acronym: HABIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Andrew Gordon, Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11204
Record Dates: First submitted 2011-08-08; First posted 2011-08-10 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Hemiplegia; Cerebral Palsy; Children
Keywords: cerebral palsy; constraint-induced therapy; constraint-induced movement therapy; CP; hemiplegia; hand; forced use; motor control; children; HABIT; Hand-arm bimanual intensive therapy; bilateral training; bimanual training; functional therapy; physical therapy; occupational therapy; intensive; pediatric; development; upper extremity; hemiplegic; childhood stroke
MeSH Terms: conditions — Hemiplegia; Cerebral Palsy; Habits | interventions — Constraint Induced Movement Therapy; Occupational Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HABIT (Experimental): Hand-Arm Bimanual Intensive Therapy (HABIT)
  Interventions: Behavioral: HABIT
- Ongoing usual and customary rehabilitation care (No Intervention): Subjects are tested over 6 months while receiving their ongoing usual and customary care schedule of physical and occupational therapy or following constraint-induced movement therapy received as usual and customary care independent of the study, and then are crossed-over to receive HABIT.

INTERVENTIONS:
Behavioral: HABIT — 90 hours of bimanual training over 3 weeks in a day camp environment
  Other Names: constraint-induced movement therapy, bimanual training, occupational therapy, physical therapy
  Arms: HABIT

SUMMARY:
A randomized control trial of bimanual training in children with hemiplegia. The protocols have been developed at Columbia University to be child friendly and draws upon our experience since 1997 with constraint-induced movement therapy in children with cerebral palsy. The investigators will test the hypothesis that bimanual training (HABIT) will result in improved hand function in children with hemiplegia.

DETAILED DESCRIPTION:
A new treatment involving bimanual (Hand-Arm Bimanual Intensive Therapy (HABIT). The protocols have been developed at Columbia University to be child friendly and draws upon our experience since 1997 with constraint-induced movement therapy in children with cerebral palsy. The investigators developed HABIT in 2004 as an alternative to constraint-therapy that avoids use of a restraint. The interventions are performed in a 15 day day-camp setting with several children and at least one therapist per child. The investigators have conducted 24 day camps to date since 2002, and are now collaborating with clinicians worldwide to expand our treatment availability. The aim is to promote the use of and improve the coordination of movement of both hands together. PARTICIPATION IS FREE. Please check out our website for more information: http://www.tc.edu/centers/cit/

ELIGIBILITY:
Inclusion Criteria:

*willingness to agree to intervention and testing procedures and travel to the University for participation and testing

Exclusion Criteria:

* health problems not associated with CP
* uncontrollable seizures
* visual problems that would interfere with carrying out the intervention or testing
* botulinum toxin therapy in the upper extremity musculature during the last six months or who wish to receive it within the period of study

Ages: 18 Months to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in quality of bimanual hand use at 12 months | 12 months
  Changes in quality of how the two hands are used during manual activity as determined from video analysis.
Change from baseline in manual dexterity at 12 months | 12 months
  Change from baseline in timed performance of standardized manual activities

SECONDARY OUTCOMES:
Change from baseline in upper extremity strength at 12 months | 12 months
Change from baseline in range of upper extremity motion at 12 months | 12 months
Change from baseline in goal achievement at 12 months | 12 months
  Change in caregiver ratings of activities identified as important goals by the caregiver

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Gordon, PhD, Principal Investigator — Teachers College, Columbia University
Locations (1):
- Teachers College, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hung YC, Casertano L, Hillman A, Gordon AM. The effect of intensive bimanual training on coordination of the hands in children with congenital hemiplegia. Res Dev Disabil. 2011 Nov-Dec;32(6):2724-31. doi: 10.1016/j.ridd.2011.05.038. Epub 2011 Jun 28. PMID 21715141
- [Background] Gordon AM, Hung YC, Brandao M, Ferre CL, Kuo HC, Friel K, Petra E, Chinnan A, Charles JR. Bimanual training and constraint-induced movement therapy in children with hemiplegic cerebral palsy: a randomized trial. Neurorehabil Neural Repair. 2011 Oct;25(8):692-702. doi: 10.1177/1545968311402508. Epub 2011 Jun 23. PMID 21700924
- [Background] Gordon AM, Schneider JA, Chinnan A, Charles JR. Efficacy of a hand-arm bimanual intensive therapy (HABIT) in children with hemiplegic cerebral palsy: a randomized control trial. Dev Med Child Neurol. 2007 Nov;49(11):830-8. doi: 10.1111/j.1469-8749.2007.00830.x. PMID 17979861
- [Background] Charles J, Gordon AM. Development of hand-arm bimanual intensive training (HABIT) for improving bimanual coordination in children with hemiplegic cerebral palsy. Dev Med Child Neurol. 2006 Nov;48(11):931-6. doi: 10.1017/S0012162206002039. PMID 17044964
- [Background] Gordon AM, Chinnan A, Gill S, Petra E, Hung YC, Charles J. Both constraint-induced movement therapy and bimanual training lead to improved performance of upper extremity function in children with hemiplegia. Dev Med Child Neurol. 2008 Dec;50(12):957-8. doi: 10.1111/j.1469-8749.2008.03166.x. No abstract available. PMID 19160464
- [Background] Gordon AM. Two hands are better than one: bimanual skill development in children with hemiplegic cerebral palsy. Dev Med Child Neurol. 2010 Apr;52(4):315-6. doi: 10.1111/j.1469-8749.2009.03390.x. Epub 2009 Oct 7. No abstract available. PMID 19811524
- See also: Center for Cerebral Palsy Research, TC, Columbia University — http://www.tc.edu/centers/cit/